CLINICAL TRIAL: NCT00023660
Title: A Phase I/II Study Of COX-2 Inhibitor, CELEBREX (CELECOXIB), And Chemoradiation In Patients With Locally Advanced Cervical Cancer
Brief Title: Radiation Therapy Plus Celecoxib, Fluorouracil, and Cisplatin in Patients With Locally Advanced Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-C-0128; CDR0000068849
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Celecoxib; Cisplatin; Fluorouracil; Brachytherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib
Drug: cisplatin
Drug: fluorouracil
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving radiation therapy in different ways and combining it with chemotherapy may kill more tumor cells. Celecoxib may slow the growth of cervical cancer by stopping blood flow to the tumor.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy plus celecoxib, fluorouracil, and cisplatin in treating patients who have locally advanced cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine treatment-related toxicity rates in patients with locally advanced cervical cancer treated with external beam radiotherapy and brachytherapy concurrently with celecoxib, fluorouracil, and cisplatin.
* Determine whether this regimen increases locoregional control rates, distant control, disease-free survival, and overall survival in these patients.
* Determine whether first-failure patterns in patients treated with this regimen are changed compared to historical controls.

OUTLINE: This is a multicenter study.

Patients undergo external beam pelvic radiotherapy once daily five days a weeks for 5 weeks beginning on day 1. Within 8 weeks, patients undergo low-dose or high-dose brachytherapy. Patients also receive concurrent chemotherapy comprising fluorouracil IV continuously over days 2-5, 23-26, and 44-47 and cisplatin IV over 4 hours on days 1, 22, and 43. Oral celecoxib is administered twice daily beginning on day 1 and continuing for 12 months.

Patients are followed every 3 months for 2 years, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 83 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous, adenocarcinoma, or adenosquamous carcinoma of the cervix

  * Stage IIB-IVA OR
  * Stage IB-IIA with pelvic node metastases and/or tumor size at least 5 cm
* No small cell, carcinoid, glassy cell, clear cell, or adenoid cystic disease
* No metastatic disease outside of pelvis
* No para-aortic disease

PATIENT CHARACTERISTICS:

Age:

* 18 to 85

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST or ALT no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 50 mL/min
* Calcium no greater than 1.3 times ULN

Cardiovascular:

* No severe heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* HIV negative
* No prior allergy to sulfonamides or non-steroidal anti-inflammatory drugs (NSAIDs)
* No prior hypersensitivity to celecoxib or any component of its formulation
* No medical or psychiatric illness that would preclude study
* No active gastrointestinal (GI) ulcer, GI bleeding, or inflammatory bowel disease
* No other prior malignancy within the past 5 years except cutaneous basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No recent prior celecoxib or other cyclo-oxygenase-2 inhibitor

Chemotherapy:

* No prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to pelvis except transvaginal radiotherapy to control bleeding

Surgery:

* No prior surgery for cervical cancer except biopsy

Other:

* No concurrent phenytoin or lithium
* No other concurrent NSAIDs

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-08; Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K. Gaffney, MD, PhD, Study Chair — University of Utah
Locations (36):
- United States (36):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mills-Peninsula Health Services, Burlingame, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - Baptist Hospital of Miami, Miami, Florida
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Ball Memorial Hospital Cancer Center, Muncie, Indiana
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital, Mount Holly, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital - Summa Health System, Akron, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Background] Viswanathan AN, Moughan J, Small W Jr, Levenback C, Iyer R, Hymes S, Dicker AP, Miller B, Erickson B, Gaffney DK. The quality of cervical cancer brachytherapy implantation and the impact on local recurrence and disease-free survival in radiation therapy oncology group prospective trials 0116 and 0128. Int J Gynecol Cancer. 2012 Jan;22(1):123-31. doi: 10.1097/IGC.0b013e31823ae3c9. PMID 22193645
- [Result] Weidhaas JB, Li SX, Winter K, Ryu J, Jhingran A, Miller B, Dicker AP, Gaffney D. Changes in gene expression predicting local control in cervical cancer: results from Radiation Therapy Oncology Group 0128. Clin Cancer Res. 2009 Jun 15;15(12):4199-206. doi: 10.1158/1078-0432.CCR-08-2257. Epub 2009 Jun 9. PMID 19509178
- [Result] Zempolich K, Fuhrman C, Milash B, Flinner R, Greven K, Ryu J, Forbes A, Kerlin K, Nichols RC, Gaffney DK. Changes in gene expression induced by chemoradiation in advanced cervical carcinoma: a microarray study of RTOG C-0128. Gynecol Oncol. 2008 May;109(2):275-9. doi: 10.1016/j.ygyno.2008.01.027. Epub 2008 Mar 4. PMID 18299147
- [Result] Gaffney DK, Winter K, Dicker AP, Miller B, Eifel PJ, Ryu J, Avizonis V, Fromm M, Greven K. A Phase II study of acute toxicity for Celebrex (celecoxib) and chemoradiation in patients with locally advanced cervical cancer: primary endpoint analysis of RTOG 0128. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):104-9. doi: 10.1016/j.ijrobp.2006.08.002. Epub 2006 Nov 2. PMID 17084549
- [Result] Gaffney DK, Winter K, Dicker AP, Miller B, Eifel PJ, Ryu J, Avizonis V, Fromm M, Small W, Greven K. Efficacy and patterns of failure for locally advanced cancer of the cervix treated with celebrex (celecoxib) and chemoradiotherapy in RTOG 0128. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):111-7. doi: 10.1016/j.ijrobp.2007.02.050. Epub 2007 May 4. PMID 17482376
- [Result] Gaffney DK, Winter K, Fuhrman C, Flinner R, Greven K, Ryu J, Forbes A, Kerlin K, Nichols RC, Zempolich K. Feasibility of RNA collection for micro-array gene expression analysis in the treatment of cervical carcinoma: a scientific correlate of RTOG C-0128. Gynecol Oncol. 2005 May;97(2):607-11. doi: 10.1016/j.ygyno.2005.01.014. PMID 15863167